CLINICAL TRIAL: NCT06935084
Title: Conducting a Randomized Controlled Trial for A Novel Patient-Facing Mobile Platform to Collect and Implement Patient-Reported Outcomes and Voice Biomarkers in Underserved Adult Patients With Asthma
Brief Title: ASTHMAXcel Voice Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Yeshiva University (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-16587
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: Mobile Health Application; Asthma Management; Asthma Control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio into one of two arms: ASTHMAXcel Voice or Usual Care (UC) arms. Block randomization (block size: 10) will be used for the purpose of balancing arms within each block. The randomization scheme will be prepared by the study statistician who will not be on study site.
Masking Description: Research assistants who administer questionnaires via the Electronic Data Capture (EDC) system will be blinded. Outcomes Assessors will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASTHMAXcel (Experimental): Participants in this arm will be provided with the adapted and refined ASTHMAXcel Voice platform.
  Interventions: Other: ASTHMAXcel Voice platform
- Usual Care (UC) (No Intervention): Participants in this arm will receive standard care.

INTERVENTIONS:
Other: ASTHMAXcel Voice platform — ASTHMAXcel Voice is a mobile health application with a multi-level approach to address barriers with intervention components and facilitate health behavior change through the use of push notifications and interactive educational content.
  Arms: ASTHMAXcel

SUMMARY:
The objective of this study is to conduct a randomized controlled trial (RCT) to compare the adapted and refined ASTHMAXcel Voice platform to usual care (UC). It is hypothesized by the investigator team that ASTHMAXcel Voice will be associated with improved clinical and process outcomes, asthma quality of life (QOL), medication adherence, and self-efficacy as compared to UC.

DETAILED DESCRIPTION:
Poor outcomes for minority patients with asthma have been linked to poverty and other social determinants of health (SDOH), environmental exposures, and poor self-management. In a previous Agency for Healthcare Research and Quality (AHRQ)-funded study, the researchers developed and pilot tested ASTHMAXcel PRO, a mobile app that promotes self-management of asthma (NCT03847142). The app was optimized for outpatient settings and promoted asthma self-management through the collection of patient-reported outcomes (PROs), animated videos, goal setting, personalized algorithms, and push notifications. The use of the app led to significant decreases in the need for steroids, visits for asthma to the emergency department, and hospitalizations for asthma.

In this current research, ASTHMAXcel Voice, an app developed and refined during enhancement of ASTHMAXcel PRO, will make use of voice biomarkers to detect worsening symptoms. This technology uses machine learning to assess respiratory dysfunction, including asthma, based on a 6-second voice sample. From the sample, a Respiratory Symptoms Risk Score (RSRS) is calculated that correlates with the speaker's risk of respiratory impairment. The updated platform will calculate the patient's RSRS; facilitate shared decision making, screen for SDoH, and referrals; improve the ability of patients to self-manage; and allow for remote care coordination.

This program draws upon the Common Sense Model (CSM) of Self-Regulation which describes a cognitive processing system that includes situational stimuli (asthma symptoms), objective representation of the health threat (illness representations) with its treatment decision (controller medication use), and appraisal of outcomes (asthma control) for the success/failure of those treatment decisions. The model contains a feedback loop with illness representations changing over time as patients gain experience with asthma management. Social Determinants of Health (SDoH) may also affect the representation of the health threat, treatment decisions, and appraisal of outcomes. As an example, a patient with depression, a poor social support network, insecure housing, and financial stress may view asthma as an acute disease that is uncontrollable, which in turn leads to negative beliefs about medications and low self-efficacy towards asthma management. ASTHMAXcel Voice strives to shift illness representations away from the belief that asthma only exists when there are active symptoms and change behavior towards daily controller medication use over the long term to prevent asthma symptoms. Realtime feedback based on voice samples that yield a RSRS (voice biomarker) will help the patient to accurately detect perceived threats and manage asthma exacerbations during earlier stages. ASTHMAXcel Voice is also based on the SEM that addresses causes of poor asthma control across four interconnected domains: community, medical system, interpersonal, and individual level factors. ASTHMAXcel Voice is a multilevel approach to address these barriers with intervention components that are directly applied at each level.

There is growing recognition that mobile health interventions can be applied across all these levels to facilitate health behavior change through the use of push notifications and interactive educational content. ASTHMAXcel Voice works on the individual and interpersonal levels by providing targeted asthma education and push notifications to assist with medication adherence and asthma management. Worse outcomes assessed by PROs (asthma control) and voice biomarkers may heighten the perceived threat level of asthma and prompt Just-in-Time Adaptive Interventions (JITAIs) to seek out the educational content more frequently to improve asthma control. On the organizational (medical system) level, ASTHMAXcel Voice will facilitate shared decision-making and ongoing communication between the patient, Community Health Worker (CHW) or Social Worker (SW), and Health Care Provider (HCP). For example, a monthly visual dashboard display will increase HCP awareness of deteriorating trends assessed from PROs and voice biomarkers. On the community level, the CHW or SW will provide patients with SDoH relevant community resources (e.g., pest remediation services, smoking cessation programs, support groups, food pantries) to address SDoH concerns reported in the mobile platform. Finally, to inform more effective design and implementation of ASTHMAXcel Voice, the study team will use the Unified Theory of Acceptance and use of Technology (UTAUT) health IT framework in determining a user's technology acceptance and adoption behavior.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Persistent asthma (diagnosed by a healthcare provider) on a daily controller medication
* Able to provide informed consent
* Smartphone access (iOS or Android) with data plan

Exclusion Criteria:

* Pregnancy
* Severe psychiatric or cognitive problems that would prohibit completion of protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control | Change from Baseline to 6 months after randomization
  Change in asthma control will be assessed and measured using the Asthma Control Test (ACT). The ACT is a 5-item questionnaire administered to assess asthma control. Participants will score each item on the ACT based on a 5-point Likert scale ranging from 1 (poor control) to 5 (excellent control) yielding an overall possible scoring range of 5-25, such that higher overall scores are associated with increased levels of asthma control. Change in ACT scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will also be used to compare ACT scores between baseline and 2 months and baseline and 6 months within each arm.

SECONDARY OUTCOMES:
Change in Asthma Control | Change from Baseline to 2 months after randomization
  Change in asthma control will be assessed and measured using the Asthma Control Test (ACT). The ACT is a 5-item questionnaire administered to assess asthma control. Participants will score each item on the ACT based on a 5-point Likert scale ranging from 1 (poor control) to 5 (excellent control) yielding an overall possible scoring range of 5-25, such that higher overall scores are associated with increased levels of asthma control. Change in ACT scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will also be used to compare ACT scores between baseline and 2 months and baseline and 6 months within each arm.
Change in User Acceptance of ASTHMAXcel Voice Application | Baseline, 2 months, and 6 months after randomization
  Change in user acceptance of the application will be assessed using the Unified Theory of Acceptance and User of Technology (UTAUT) Questionnaire. The UTAUT considers 4 constructs: performance expectancy (PE), effort expectancy (EE), social influence (SI), and facilitating conditions (FC), as most influential in determining technology acceptance and adoption behavior. Each of the 4 constructs consists of 4 statements which are evaluated on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree), with higher scores indicating a greater likelihood of technology acceptance and use, reflecting stronger perceptions of PE, EE, SI, and FC. Scores for all items are summed and then the total score is divided by 16 to calculate a mean or average score. Scores will be summarized by using basic descriptive statistics. Paired t-tests will also be used to assess changes in user acceptance between baseline and 2 months and baseline and 6 months within the arm.
Change in User Satisfaction of Interaction with the ASTHMAXcel Voice application | Baseline, 2 months, and 6 months after randomization
  Change in User satisfaction of Interaction with the application will be assessed using Version 7 of the Questionnaire for User Interface Satisfaction (QUIS). The QUIS is a measurement tool designed to assess a computer user's subjective satisfaction with specific aspects of the human-computer interface. QUIS measures specific interface factors such as screen visibility, terminology and system information, learning factors, system capabilities, usability and user interface, and system clutter, across 32 questions. Each QUIS question is measured on an ascending scale ranging from 0-9, wherein higher scores are associated with more favorable user impression of aspects of the interface. Scores for all items are summed and divided by the number of items answered to calculate a mean or average score. Scores will be summarized by using basic descriptive statistics. Paired t-tests will also be used to assess changes between baseline and 2 months and baseline and 6 months within the arm.
ASTHMAXcel Voice application Usage | 2 months and 6 months after randomization
  ASTHMAXcel Voice application usage will be evaluated using analytics within the "Admin Panel" of the application. Specifically, the number of logins to ASTHMAXcel Voice will be determined and considered as a proxy for usage. Usage will be summarized using basic descriptive statistics.
Change in Overall User Satisfaction | Baseline, 2 months, and 6 months after randomization
  Overall User Satisfaction will be assessed using the 8-item Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is a brief global measure of client satisfaction which contains four response choices (1-4), where "1" indicates the lowest degree of satisfaction and "4," the highest. Scores are summed across each item once. Responses to items 2, 4, 5, and 8 are reverse scored. Total overall scores range from 8-32, where in higher scores are indicative of greater overall user satisfaction. Scores will be summarized by using basic descriptive statistics. Paired t-tests will also be used to assess changes between post-refinement baseline and 2 months and baseline and 6 months within the arm.
Change in Shared Decision Making | Baseline to 2 months and 6 months after randomization
  Patient-reported degree of shared decision making will be assessed using the 9-item Shared Decision-Making Questionnaire (SDM-Q-9). The SDM-Q-9 consists of 9 statements which asks the patient to assess the extent to which they agree or disagree with elements and perceptions of shared decision-making during clinical encounters. Each statement on the SDM-Q-9 is scored on a 6-point Likert scale ranging from 0 (completely disagree) to 5 (completely agree). Scores are summed to yield an overall possible scoring range of 0-45, with higher values being indicative of greater perceived shared decision making. Scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will also be used to assess changes between post-refinement baseline and 2 months and 6 months within the arm
Change in Asthma-related Quality of Life | Baseline to 2 months and 6 months after randomization
  Change in Asthma-related Quality of Life will be assessed using the Mini Asthma Quality of Life Questionnaire (MiniAQLQ). The MiniAQLQ is a 15-item questionnaire that assesses asthma-related quality of life. Participants are asked to evaluate each of the questions/statements to describe how much (relative) time has been spent attending to symptoms of asthma or how much asthma has limited activities over the past 2 weeks. Each of the 15 items is scored on a 7-point Likert scale ranging from 1 (severe impairment) to 7 (no impairment), such that higher scores are associated with a better overall quality of life. Scores for the 15-items are summed and divided by 15 to express as a score out of 7 (mean or average score). Change in asthma quality of life scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will also be used to assess changes in asthma-related quality of life between baseline and 2 months and baseline and 6 months within each arm.
Asthma Healthcare Utilization - Emergency Department (ED) Visits | 2 months and 6 months after randomization
  The number of asthma-related ED visits at 2 months and 6-months post-randomization will be summarized by study arm using basic descriptive statistics.
Asthma Healthcare Utilization - Hospitalizations | 2 months and 6 months after randomization
  The number of asthma-related hospitalizations at 2 months and 6-months post-randomization will be summarized by study arm using basic descriptive statistics.
Change in Self-efficacy for managing chronic diseases | Baseline to 2 months and 6 months after randomization
  Self-efficacy for managing chronic diseases will be evaluated using the Self-Efficacy for Managing Chronic Disease 6-Item (SEMCD-6) Scale. The SEMCD-6 assesses the level of confidence in managing six areas related to chronic disease: fatigue, physical discomfort/pain, emotional distress, other symptoms/health problems, tasks/activities needed to manage health conditions, and things other than just taking medication. Each question is rated on a 10-point scale ranging from 1 (not confident at all) to 10 (totally confident). Scores for all six items are summed, and then the total score is divided by six to calculate a mean or average score. Higher scores are associated with greater self-efficacy. Group scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will also be used to assess changes between post-refinement baseline and 2 months and 6 months within the arm.
Change in Self-reported Medication Adherence | Baseline to 2 months and 6 months after randomization
  Medication Adherence will be evaluated using the 5-Item Medication Adherence Report Scale (MARS-5). The MARS-5 is a self-reported tool used to assess medication adherence and consists of 5 questions including items related to forgetting, changing dosage, stopping, skipping, and taking less medication. Each question is answered on a 5-point Likert scale (1=always, 2=often, 3=sometimes, 4=rarely, and 5=never), resulting in an overall possible score of 5-25, with higher scores indicating a higher level of adherence. Group scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will also be used to assess changes between post-refinement baseline and 2 months and 6 months within the arm
SDoH Screening | 2 months and 6 months after randomization
  SDoH Screening will be determined by the number of SDoH positive screens over the prior month. Group scores will be summarized by study arm using basic descriptive statistics.
SDoH Referral | 2 months and 6 months after randomization
  SDoH Referral will be determined by the number of completed SDoH referrals over the prior month. Group scores will be summarized by study arm using basic descriptive statistics.
Referral Completion Rate | 2 months and 6 months after randomization
  SDoH Referral Completion Rate will be assessed by the number of SDoH referral completions over the prior month. Group scores will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Jariwala, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Once primary study findings have been published, deidentified data publicly available along with its associated documentation. Public Use Data: All de-identified study data that are not designed as restricted use will be made publicly available as supplementary material of articles in PubMed Central. All datasets will require detailed metadata documentation (Word documents), including (but not limited to) the methodology and procedures used to collect the data, details about codes (codebooks), definitions of variables, variable field locations, frequencies, etc. All data sets that are shared will be accompanied by the relevant metadata. No other specialized tools will be needed to access or manipulate shared scientific data to support replication or reuse.
  Participant-level data from this study will be fully de-identified and represented as an OMOP-CDM v5.3.1 dataset (mapped to OHDSI/Athena vocabulary system)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Results generated from this grant will be presented at national or international scientific meetings and conferences and will be published in a timely fashion. Data sets and associated documents will be provided to the NIH study Program Official within timelines described in the NIH Policy for Data Sharing from Observational Epidemiology Studies - no later than 3 years after the completion of each examination or follow-up cycle or 2 years after the baseline, follow-up, genetic, ancillary study, or other data set is finalized within the study for analysis for use in publication, whichever comes first. Study data will be made available to other users after publication of the study's main results have been published (estimated to be within 12 months of study closure). Once available, no time limit will be placed on accessibility of the study data.

REFERENCES:
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] Chan AHY, Horne R, Hankins M, Chisari C. The Medication Adherence Report Scale: A measurement tool for eliciting patients' reports of nonadherence. Br J Clin Pharmacol. 2020 Jul;86(7):1281-1288. doi: 10.1111/bcp.14193. Epub 2020 May 18. PMID 31823381
- [Background] Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014 Nov;67(11):1265-73. doi: 10.1016/j.jclinepi.2014.06.009. Epub 2014 Aug 3. PMID 25091546
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Leventhal H, Brissette, I., Leventhal, E. A. The common sense model of self-regulation of health and illness. In: Cameron LD, Leventhal, H., ed. The self-regulation of health and illness behavior. London, UK: Taylor and Francis Books; 2003:42-65.
- [Background] Sofianou A, Martynenko M, Wolf MS, Wisnivesky JP, Krauskopf K, Wilson EA, Goel MS, Leventhal H, Halm EA, Federman AD. Asthma beliefs are associated with medication adherence in older asthmatics. J Gen Intern Med. 2013 Jan;28(1):67-73. doi: 10.1007/s11606-012-2160-z. Epub 2012 Aug 10. PMID 22878848
- [Background] Arcoleo KJ, McGovern C, Kaur K, Halterman JS, Mammen J, Crean H, Rastogi D, Feldman JM. Longitudinal Patterns of Mexican and Puerto Rican Children's Asthma Controller Medication Adherence and Acute Healthcare Use. Ann Am Thorac Soc. 2019 Jun;16(6):715-723. doi: 10.1513/AnnalsATS.201807-462OC. PMID 30860858
- [Background] U B. Toward an experimental ecology of human development. American Psychologist. 1977;32(7):513 531.
- [Background] Kolff CA, Scott VP, Stockwell MS. The use of technology to promote vaccination: A social ecological model based framework. Hum Vaccin Immunother. 2018 Jul 3;14(7):1636-1646. doi: 10.1080/21645515.2018.1477458. Epub 2018 Jul 3. PMID 29781750
- [Background] Venkatesh V MM, Davis GB, Davis FD. User acceptance of information technology: Toward a unified view. MIS quarterly. 2003;1:425-478.
- [Background] U.S. Department of Health and Human Services NIoH. Expert Panel Report 3: Guidelines for the Diagnosis and Management of Asthma (EPR-3). 2007 Jul.
- [Background] Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009 Oct;124(4):719-23.e1. doi: 10.1016/j.jaci.2009.06.053. Epub 2009 Sep 19. PMID 19767070
- [Background] Hsia BC, Wu S, Mowrey WB, Jariwala SP. Evaluating the ASTHMAXcel Mobile Application Regarding Asthma Knowledge and Clinical Outcomes. Respir Care. 2020 Aug;65(8):1112-1119. doi: 10.4187/respcare.07550. Epub 2020 Jun 2. PMID 32487751
- [Background] Hanson JL, Balmer DF, Giardino AP. Qualitative research methods for medical educators. Acad Pediatr. 2011 Sep-Oct;11(5):375-86. doi: 10.1016/j.acap.2011.05.001. Epub 2011 Jul 23. PMID 21783450
- [Background] Hsia B, Mowrey W, Keskin T, Wu S, Aita R, Kwak L, Ferastraoarou D, Rosenstreich D, Jariwala SP. Developing and pilot testing ASTHMAXcel, a mobile app for adults with asthma. J Asthma. 2021 Jun;58(6):834-847. doi: 10.1080/02770903.2020.1728770. Epub 2020 Feb 19. PMID 32046564
- [Background] Figueroa JF, Frakt AB, Jha AK. Addressing Social Determinants of Health: Time for a Polysocial Risk Score. JAMA. 2020 Apr 28;323(16):1553-1554. doi: 10.1001/jama.2020.2436. No abstract available. PMID 32242887